CLINICAL TRIAL: NCT06756646
Title: Exploring the Effects of Aerobic Exercise Combined with Blood Flow Restriction Training on Exercise Capacity, Cardiopulmonary Functions, and Quality of Life in Patients with Chronic Obstructive Pulmonary Disease
Brief Title: Exploring the Effects of Aerobic Exercise Combined with BFRT on Patients with COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Kun-Ling Tsai, Professor and Chair, Department of Physical Therapy, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B-ER-113-298
Record Dates: First submitted 2024-12-19; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Blood flow restriction training; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual care group (Active Comparator): The Usual care group will receive COPD and exercise-related education.
  Interventions: Behavioral: Disease and exercise suggestion
- Aerobic exercise group-cycling (Experimental): The aerobic exercise group will receive cycling training intervention 2-3 times per week for 2 months.
  Interventions: Behavioral: Aerobic exercise intervention
- BFR group-cycling + BFR (Experimental): The BFR group will receive cycling training combined with BFR intervention 2-3 times per week for 2 months.
  Interventions: Behavioral: Blood flow restriction (BFR) intervention

INTERVENTIONS:
Behavioral: Aerobic exercise intervention — The aerobic exercise intervention will utilize an ergometer. The program will be conducted 2-3 times per week over a 3-month period.
  Arms: Aerobic exercise group-cycling
Behavioral: Disease and exercise suggestion — The participants will be provided by educational program about COPD self-care and home-based exercise approach.
  Arms: Usual care group
Behavioral: Blood flow restriction (BFR) intervention — Blood flow restriction (BFR) intervention will combine aerobic exercise on the ergometer with BFR training. The program will be conducted 2-3 times per week over a 3-month period.
  Arms: BFR group-cycling + BFR

SUMMARY:
Investigate the effects of exercise training on the cardiopulmonary function and exercise capacity in COPD patients.

DETAILED DESCRIPTION:
The systemic effects of Chronic Obstructive Pulmonary Disease (COPD) can precipitate a series of complications, including cardiovascular disorders, muscle atrophy, and osteoporosis. These comorbid conditions often result in decreased physical activity and suboptimal physical fitness, compelling patients to lead a sedentary lifestyle to mitigate exercise-induced dyspnea. Addressing the limitations in exercise tolerance remains a critical therapeutic goal in the treatment of COPD. According to research, exercise intolerance is caused by both poor pulmonary function and associated skeletal muscle dysfunction. Blood flow restriction training, a new rehabilitation technique, has shown promise in improving muscular strength at lower exercise intensities and in shorter timeframes, presenting a fresh approach to COPD rehabilitation.

The research aims to investigate the impact of incorporating blood flow restriction training into a holistic aerobic exercise program on exercise capacity and quality of life among patients with COPD. The findings are intended to clarify the potential of this innovative training technique as a supplementary therapeutic strategy in the management of COPD.

ELIGIBILITY:
Inclusion Criteria:

1. COPD classified as levels 2-4.
2. Stable condition without worsening in the past three months.
3. No participation in any rehabilitation program within the past six months.
4. Ability to understand and follow verbal commands and cooperate with an exercise training program.

Exclusion Criteria:

1. Unconscious or unable to cooperate with the evaluator.
2. Hospitalization due to acute illness within the past three months.
3. Severe joint diseases or history of lower limb surgery.
4. Severe cardiovascular disease (e.g., presence of a cardiac pacemaker or acute myocardial infarction within the past six months).
5. Dependence on oxygen supply.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxygen consumption (VO2) | Change from baseline (0 week) to follow up (20 weeks)
  Oxygen consumption examined by cardiopulmonary exercise test
Diaphragm capacity | Change from baseline (0 week) to follow up (20 weeks)
  Diaphragm capacity examined by diaphragmatic ultrasound

SECONDARY OUTCOMES:
Functional capacity | Change from baseline (0 week) to follow up (20 weeks)
  Functional capacity examined by 6MWT
Heart Rate Variability | Change from baseline (0 week) to follow up (20 weeks)
  Heart Rate Variability examined by autonomic nervous system
Pulmonary function test | Change from baseline (0 week) to follow up (20 weeks)
  Pulmonary function test examined by spirometer. Spirometry is a physiological test that measures the ability to inhale and exhale air over time. The main spirometry results are forced vital capacity (FVC), forced expiratory volume in the first second (FEV1), and the FEV1/FVC ratio.
Maximum respiratory pressure | Change from baseline (0 week) to follow up (20 weeks)
  Maximum respiratory pressure examined by pressure meter
Quality of life score (COPD-related questionnaire-I) | Change from baseline (0 week) to follow up (20 weeks)
  Quality of life score examined by mMRC Questionnaire.
Quality of life score (COPD-related questionnaire-II) | Change from baseline (0 week) to follow up (20 weeks)
  COPD Assessment Test (CAT) questionaire
Quality of life score (COPD-related questionnaire-III) | Change from baseline (0 week) to follow up (20 weeks)
  St George's Respiratory Questionnaire (SGRQ)

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ling Tsai, Ph.D., Principal Investigator — Department of Physical Therapy, National Cheng Kung University
Locations (1):
- National Cheng Kung University Hostipal, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD sharing plan will be decided after summarized data being published.